CLINICAL TRIAL: NCT06053333
Title: Social Determinants of Health in Hepatobiliary Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-012368; NCI-2023-05784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-012368 (Other: Mayo Clinic in Rochester); K23MD017217 (NIH)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Malignant Hepatobiliary Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete a questionnaire, undergo blood, urine, and buccal swab sample collection and have their medical records reviewed on study. Patients also undergo collection of clinically archived tissue samples on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates barriers to receiving care and risks associated with developing cancer among patients diagnosed with hepatobiliary cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize the social determinants of health - and specifically travel-limiting access to cancer care but also other issues, such as trouble in finding childcare, joblessness, and limited education - among SEA Americans with hepatobiliary cancers, exposure risk including aflatoxin and viral hepatitis among other exposures.

OUTLINE: This is an observational study.

Patients complete a questionnaire, undergo blood, urine, and buccal swab sample collection and have their medical records reviewed on study. Patients also undergo collection of clinically archived tissue samples on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18+ year of age with hepatobiliary cancers

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with hepatobiliary cancers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2028-07-17 (Estimated); Study Completion 2028-07-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients reporting transportation barriers that affect medical care | Baseline; up to 2 years
  Estimated using Social Determinants of Health Screening Tool designed by the American Academy of Family Medicine, by the proportion of patients who respond "yes" to the question, "Do you put off or neglect going to the doctor because of distance or transportation?".

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen H. Tran, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials